CLINICAL TRIAL: NCT05018273
Title: A Phase 1B, Open-Label, Dose-Escalation Study of the Safety of and Antigen-specific Immune Responses Elicited by VB10.NEO in Combination With Atezolizumab in Patients With Locally Advanced and Metastatic Tumors
Brief Title: Study of VB10.NEO in Combination With Atezolizumab in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nykode Therapeutics ASA (Industry)
Collaborators: Genentech, Inc. (Industry); Vaccibody AS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB N-02
Record Dates: First submitted 2021-07-13; First posted 2021-08-24 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumors, Adult
Keywords: Locally advanced and metastatic tumors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VB10.NEO 3 mg in combination with Atezolizumab 1200 mg (Experimental): VB10.NEO 3 mg will be administered by IM injection for an induction course Q3W (4 doses) followed by maintenance doses Q6W (6 doses) and Q12W (5 doses).
  Atezolizumab 1200 mg will be administered by intravenous (IV) infusion on Day 1 of 21 day cycles.
  Interventions: Biological: VB10.NEO
- VB10.NEO 6 mg in combination with Atezolizumab 1200 mg (Experimental): VB10.NEO 6 mg will be administered by IM injection for an induction course Q3W (4 doses) followed by maintenance doses Q6W (6 doses) and Q12W (5 doses).
  Atezolizumab 1200 mg will be administered by intravenous (IV) infusion on Day 1 of 21 day cycles.
  Interventions: Biological: VB10.NEO
- VB10.NEO 9 mg in combination with Atezolizumab 1200 mg (Experimental): VB10.NEO 9 mg will be administered by IM injection for an induction course Q3W (4 doses) followed by maintenance doses Q6W (6 doses) and Q12W (5 doses).
  Atezolizumab 1200 mg will be administered by intravenous (IV) infusion on Day 1 of 21 day cycles.
  Interventions: Biological: VB10.NEO

INTERVENTIONS:
Biological: VB10.NEO — The personalized vaccine VB10.NEO vaccine is given in combination with the PD-L1 inhibitor atezolizumab.
  Other Names: Atezolizumab; Tecentriq

SUMMARY:
A phase 1b, open-label, multicenter, dose-escalation study designed to evaluate the safety, tolerability, antigen-specific immune response and preliminary antitumor activity associated with VB10.NEO administered in combination with atezolizumab, and to identify a RP2D for VB10.NEO in combination with atezolizumab, in patients with locally advanced and metastatic tumors that have progressed after at least 1 available standard therapy; or for whom standard therapy has proven to be ineffective or intolerable, or is considered inappropriate; or for whom a clinical trial of an investigational agent is a recognized standard of care (SOC).

ELIGIBILITY:
Inclusion Criteria:

Tumor types: melanoma, NSCLC, RCC, UC, HNSCC, TNBC, gastric/GEJ cancer, cervical, anal, or MSI-high tumors. Additionally up to 15 subjects with other locally advanced or metastatic solid tumor types not listed above.

Signed Informed Consent Form

Age ≥18 years at time of signing the Informed Consent Form

Ability to comply with the trial protocol

ECOG Performance Status of ≤ 1: Note: If ECOG Performance Status at Screen 2B assessment was performed > 7 days prior to VB10.NEO start date, it needs to be re-assessed on C1D1 prior to administration of VB10.NEO and remain ≤ 1

GRIm score ≤ 1 at Screen 1, this only applies for subjects initially screened under protocol version 5

Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 7 days prior to initiation of trial treatment:

ANC ≥1.5 × 109/L (1500/µL) Must be met without administration of growth factors within 2 weeks prior to treatment start date.

Lymphocyte count ≥0.5 × 109/L (500/µL)

Platelet count 100-450 × 109/L (100,000 - 450,000/µL) Must be met without administration of platelet transfusion within 2 weeks prior to treatment start date.

Hemoglobin ≥90 g/L (9 g/dL) Must be met without erythropoietin dependency and without red blood cell transfusion within 2 weeks prior to treatment start date.

AST and ALT ≤3 × ULN

Alkaline phosphatase (ALP) ≤2.5 × ULN, with the following exceptions:

Subjects with documented liver or bone metastases: ALP ≤5 × ULN

Total bilirubin ≤1.5 × ULN with the following exception:

Subjects with known Gilbert disease: total bilirubin ≤3 × ULN

Measured or calculated creatinine clearance ≥50 mL/min (according to the Cockcroft-Gault formula)

Albumin ≥25 g/L (2.5 g/dL)

For subjects not receiving therapeutic anticoagulation: International Normalized Ratio (INR) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN

For subjects receiving therapeutic anticoagulation: stable anticoagulant regimen

Female subjects of childbearing potential must have a negative serum pregnancy test result within 72 hours prior to initiation of trial treatment.

Female subjects of childbearing potential must agree to use a highly effective form of contraception during treatment and for at least 90 days after the final dose of VB10.NEO, and for 5 months after the final dose of atezolizumab, whichever occurs later. Highly effective forms of contraception include:

combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal

progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable

intrauterine device

intrauterine hormone-releasing system

bilateral tubal occlusion

vasectomized partner

sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence [calendar, symptothermal, post-ovulation methods], withdrawal [coitus interruptus], spermicides only, and the lactational amenorrhea method are not acceptable methods of contraception).

For men with a female partner of childbearing potential or pregnant female partner: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom during the treatment period and for at least 28 days after the final dose of trial treatment to avoid exposing the embryo, and agreement to refrain from donating sperm.

Exclusion Criteria:

Pregnant or breastfeeding, or intending to become pregnant during the trial or within 90 days after the last dose of VB10.NEO or 5 months after the last dose of atezolizumab, whichever occurs later

Significant cardiovascular disease such as, but not limited to, New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina

QT interval corrected through use of Fridericia's formula (QTcF) >470ms demonstrated by at least 2 electrocardiograms (ECGs) >30 minutes apart

Clinically significant liver disease including active viral, alcoholic, or other hepatitis, cirrhosis, and inherited liver disease or current alcohol abuse

Positive hepatitis B surface antigen (HBsAg) test at screening

Subjects with past or resolved hepatitis B infection (defined as having a negative HBsAg test and a positive IgG antibody to hepatitis B core antigen) are eligible.

Positive hepatitis C virus (HCV) antibody test at screening

Subjects positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)

Positive human immunodeficiency virus (HIV)-1 test at screening

Active tuberculosis

Any other diseases, metabolic dysfunction, physical examination finding, and/or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or may render the subject at high risk from treatment complications

Known primary immunodeficiencies

Active, or history of, autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

Subjects with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the trial.

Subjects with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the trial.

Subjects with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., subjects with psoriatic arthritis are excluded) are eligible for the trial provided all of the following conditions are met:

Rash must cover <10% of body surface area

Disease is well controlled at baseline and requires only low potency topical corticosteroids

No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months

History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.

Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation.

Known allergy or hypersensitivity to any component of the VB10.NEO formulation.

History of idiopathic pulmonary fibrosis, pneumonitis (including drug-induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on imaging conducted for tumor assessment at screening

History of radiation pneumonitis in the radiation field (fibrosis) is permitted

History of drug-induced pneumonitis that was asymptomatic (defined by radiographic findings only) and reversible (without any anti-inflammatory therapies) is permitted.

Severe infection within 28 days prior to Cycle 1, Day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia

Subjects receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease [COPD] exacerbation) are eligible for the trial.

Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

Subjects with indwelling catheters (e.g., PleurX) are allowed.

Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL, or corrected calcium >ULN)

Major surgical procedure within 28 days prior to Cycle 1, Day 1, or anticipation of need for a major surgical procedure during the course of the trial

Prior allogeneic stem cell or solid organ transplantation

Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 28 days or 5 drug-elimination half-lives (whichever is longer) prior to Cycle 1, Day 1

Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone >7.5 mg/day, cyclophosphamide, azathioprine, methotrexate, thalidomide, and tumor necrosis factor-alpha [TNF-α] antagonists) within 2 weeks prior to Cycle 1, Day 1 with the following exceptions:

Subjects who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the trial after medical monitor confirmation has been obtained

Subjects who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for COPD or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the trial.

Treatment with investigational therapy within 28 days prior to Cycle 1, Day 1

Live, attenuated vaccines are prohibited within 28 days prior to Cycle 1, Day 1, during atezolizumab treatment, and for 5 months after the final dose of atezolizumab

Vaccination with an approved COVID-19 vaccine that does not contain live, attenuated virus is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From baseline and up to 27 months
  The number and percentage of participants that experience an adverse event (AE)
Changes from baseline in vital signs | From baseline and up to 27 months
  Changes for measurements done prior and after the first VB10.NEO injection of each cycle for the following vital signs: Systolic blood pressure (mmHg); diastolic blood pressure (mmHg); pulse rate (bpm); respiration rate (breaths/min); body temperature (°C)
Changes from baseline in clinical laboratory parameters | From baseline and up to 27 months
  Changes for clinical laboratory parameters analysed locally prior and after the first VB10.NEO injection of each cycle, including hematology, chemistry panel, coagulation, thyroid function testing, C-reactive protein, urinalysis and serology

SECONDARY OUTCOMES:
Assessment of the antigen-specific immune response elicited by VB10.NEO administered in combination with atezolizumab | From baseline and up to 25 months
  Number and magnitude of antigen-specific T-cell responses before and after initiation of trial treatment
Objective response rate (ORR) | From baseline and up to 27 months
  The proportion of subjects with a complete response (CR) or partial response (PR) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of response (DOR) | From baseline and up to 27 months
  The time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Progression free survival (PFS) | From baseline and up to 27 months
  The time from the first trial treatment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Overall survival (OS) | From baseline and up to 27 months
  The time from the first trial treatment to death from any cause
Characterize the pharmacokinetic of atezolizumab when administered in combination with VB10.NEO. | From baseline and up to 25 months
  Serum concentration of atezolizumab at specified timepoints
Evaluate the immune response to atezolizumab when administered in combination with VB10.NEO | From baseline and up to 25 months
  Prevalence of antidrug antibodies (ADAs) to atezolizumab at baseline and incidence of ADAs to atezolizumab

OTHER OUTCOMES:
Dose finding objective | Through study completion, an average of 2 years.
  Identify a recommended phase 2 dose (RP2D) and regimen for VB10.NEO in combination with atezolizumab by evaluating the relationship between VB10.NEO dose and safety, biomarker, and antitumor activity endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Siri Torhaug, MD, Study Director — Nykode Therapeutics ASA
Locations (12):
- United States (5):
  - The Regents of the University of California, San Francisco, California
  - Yale Cancer Institute, New Haven, Connecticut
  - Norton Cancer Institute, Louisville, Kentucky
  - Washington University, St Louis, Missouri
  - MD Andersson, Houston, Texas
- Germany (2):
  - Charité-Universitätsmedizin Berlin, Berlin
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
- Spain (5):
  - Hospital Universitario Virgen de la Victoria, Campus Universitario De Teatinos s/n, Málaga, MA
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No